CLINICAL TRIAL: NCT05679401
Title: A Phase 3 Open-label, Controlled, Randomised, Multi-centre Trial Comparing Imlifidase and Standard-of-care With Standard-of-care Alone in the Treatment of Severe Anti-GBM Antibody Disease (Goodpasture Disease)
Brief Title: A Study With Imlifidase in Anti-GBM Disease
Acronym: GOOD-IDES-02
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hansa Biopharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-HMedIdeS-24; 2022-500121-33-01 (Other: EU Trial Number); 1005498 (Other: Integrated Research Application System (IRAS), UK)
Record Dates: First submitted 2022-12-15; First posted 2023-01-11 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Anti-Glomerular Basement Membrane Disease; Anti-Glomerular Basement Membrane Antibody Disease; Goodpasture Syndrome; Good Pasture Syndrome
Keywords: Anti-GBM
MeSH Terms: conditions — Anti-Glomerular Basement Membrane Disease; Rapidly progressive glomerulonephritis with pulmonary hemorrhage | interventions — Mac-1-like protein, Streptococcus; Plasma Exchange; Cyclophosphamide; Glucocorticoids

STUDY DESIGN:
Intervention Model Description: Open-label, controlled, randomised, multi-centre trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Imlifidase and Standard-of-Care (SoC) (Experimental): * Imlifidase is administered IV as one dose of 0.50 mg/kg over 30 minutes.
  * SoC consists of a standardized combination of PLEX, CYC, and glucocorticoids.
  Interventions: Drug: Imlifidase; Procedure: Plasma exchange (PLEX); Drug: Cyclophosphamide (CYC); Drug: Glucocorticoids
- Standard-of-Care (SoC) (Active Comparator): SoC consists of a standardized combination of PLEX, CYC, and glucocorticoids.
  Interventions: Procedure: Plasma exchange (PLEX); Drug: Cyclophosphamide (CYC); Drug: Glucocorticoids

INTERVENTIONS:
Drug: Imlifidase — Imlifidase is an immunoglobulin G (IgG)-degrading enzyme of Streptococcus pyogenes that is highly selective towards IgG. The cleavage of IgG generates one F(ab')2- and one homodimeric Fc-fragment and efficiently neutralizes Fc-mediated activities of IgG.
  Other Names: IdeS, HMED-IdeS
  Arms: Imlifidase and Standard-of-Care (SoC)
Procedure: Plasma exchange (PLEX) — PLEX removes the patient's pathogenic anti-GBM antibodies, by replacement of deficient plasma with a replacement fluid.
  Other Names: PE
Drug: Cyclophosphamide (CYC) — Cyclophosphamide's main mechanism of action (i.e. crosslinking of strands of DNA and RNA) results in inhibition of protein synthesis. Hence treatment prevents formation of new anti-GBM antibodies.
Drug: Glucocorticoids — Glucocorticoids inhibit the inflammation process.

SUMMARY:
An open-label, controlled, randomised, multi-centre Phase 3 trial evaluating renal function in patients with severe anti-GBM disease comparing imlifidase and standard of care (SoC) with SoC alone. All patients will remain in the trial for 24 months.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo screening to determine eligibility for study entry. Patients will be randomised to treatment in a 1:1 ratio to either imlifidase and SoC or SoC only.

SoC consists of a combination of plasma exchange (PLEX), cyclophosphamide (CYC), and glucocorticoids. For patients randomised to the imlifidase arm the first PLEX immediately after randomisation is replaced by administration of imlifidase.

Kidney function, anti-GBM antibody levels, pulmonary symptoms, safety, pharmacokinetic/pharmacodynamic (PK/PD) and health related quality of life (HRQoL) among others, will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Anti-GBM antibodies constituting an indication for PLEX as judged by the Investigator
2. Haematuria on dipstick and/or urinary sediment
3. eGFR(MDRD) <20 mL/min/1.73 m^2
4. Patients aged ≥18 years
5. Willing and able to give written Informed Consent and to comply with the requirements of the study protocol

Exclusion Criteria:

1. Diagnosis of anti-GBM disease more than 14 days prior to randomisation
2. Anuria during the last 24-hour
3. Any constituent of SoC given more than 10 days prior to randomisation
4. IVIg within 4 weeks before randomisation
5. History or presence of any medical condition or disease which, in the opinion of the investigator, may place the patient at unacceptable risk, or jeopardise the purpose of the study
6. Patients previously randomised in the study
7. Unsuitable to participate in the trial for any other reason in the opinion of the investigator
8. Pregnancy or breast feeding
9. Contraception:

   1. Men who are not vasectomised or abstinent or with a partner (of child-bearing potential) not willing to use one of the highly effective contraceptives listed below from screening to 6 months following discontinuation of CYC
   2. Men who are not willing to refrain from donating sperm from screening to 6 months following discontinuation of CYC
   3. Men who are not willing to use a condom during any form of sexual intercourse, regardless of a partner being of child-bearing potential from screening to 6 months following discontinuation of CYC
   4. Women of child-bearing potential not willing or not able to use at least one highly effective contraceptive method from screening to 12 months following discontinuation of CYC.

   In the context of this trial, a highly effective method is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly such as:
   * combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral/intravaginal/transdermal)
   * progestogen-only hormonal contraception associated with inhibition of ovulation (oral/injectable/implantable)
   * intrauterine device (IUD)
   * intrauterine hormone-releasing system (IUS)
   * bilateral tubal occlusion
   * vasectomised partner
   * true abstinence: When this is in line with the preferred and usual lifestyle of the patient. [Periodic abstinence (such as calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception]
10. Previous imlifidase treatment or known hypersensitivity to any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Renal function as evaluated by estimated glomerular filtration rate (eGFR) at 6 months | At 6 months after randomisation

SECONDARY OUTCOMES:
Proportion of patients with functioning kidney at 6 months | At 6 months after randomisation
Time to non-toxic level of anti-GBM antibodies | During the study from screening up to 6 months
Exposure to toxic level of anti-GBM antibodies | From randomisation up to Day 22 and to Day 29 respectively
  Exposure to anti-GBM antibodies will be assessed by evaluation of the area under the anti-GBM antibody concentration versus time curve.
Renal function as evaluated by eGFR at 3 months | At 3 months after randomisation
Proportion of patients with functioning kidney at 3 months, | At 3 months after randomisation
Proportion of patients experiencing end stage renal disease (ESRD) within 6 months | During the study from randomisation up to 6 months
Proportion of patients experiencing death due to anti-GBM disease within 6 months | During the study from randomisation up to 6 months
Change in urine creatinine clearance (CrCl) from randomisation to 3 and 6 months | At randomisation and at 3 and 6 months
U-albumin/creatinine ratio at 3 and 6 months (24h collection) | At screening and at 3 and 6 months
U-albumin/creatinine ratio at screening and during study (morning urine void) | During the study from screening up to 6 months
Renal function as evaluated by eGFR at screening and during study | During the study from screening up to 6 months
Number of PLEX sessions within 3 months from randomisation | During the study from randomisation up to 3 months
Number of days on dialysis within 3 and 6 months from randomisation | During the study from randomisation to 3 months and 6 months
Proportion of patients being negative during study for anti-GBM antibodies/anti-neutrophilic cytoplasmic autoantibodies (ANCA)/anti-GBM antibodies+ANCA | During the study from screening up to 6 months
Number of days with mechanical ventilation due to anti-GBM disease within 3 months from randomisation | During the study from randomisation to 3 months
Number of days at intensive care unit (ICU) and number of days in hospitalisation from randomisation to 3 months | During the study from randomisation to 3 months
Change in health related quality of life (HRQoL) from screening to 6 months | At screening and at 6 months
  All patients will fill out the HRQoL questionnaire PROMIS-29 which is a universal rather than disease specific measure.
  The PROMIS-29 measure assesses pain intensity using a single 0-10 numeric pain rating item and seven health domains using four items each: physical functioning, fatigue, pain interference, depression, anxiety, ability to participate in social roles and activities, and sleep disturbance. The score of each domain is converted into a standardized score so called T-score reported for each patient. A T-score of 50 represent a person from a reference population. A T-score higher than 50 indicates more of what is measured and a T-score less than 50 indicates less of what is measured.
Change in health status from screening to 6 months | At screening and at 6 months
  All patients will fill out the EQ-5D-5L questionnarie that comprises 5 questions measuring 5 dimensions of health status (mobility, self-care, usual activities, pain/ discomfort, and anxiety/depression). Patients will be asked to select a response to each category that best describes their current health. The EQ-5D-5L also contains a visual analogue scale and the patients will be asked to rate their health on a scale of 0-100.
Pharmacokinetic (PK) data (Cmax) from start of treatment to Day 15 | During the study from before administration of imlifidase up to Day 15
  Cmax = Maximum observed plasma concentration of imlifidase following dosing.
Imlifidase pharmacodynamic (PD) profile (IgG levels in serum) from start of treatment to Day 15 | During the study from before administration of imlifidase up to Day 15
  Imlifidase cleaves IgG. PD of imlifidase will be assessed as IgG levels in serum. A validated electrochemiluminescence (ECL) method will be used for the analysis.
Imlifidase pharmacodynamic (PD) profile (composition of different IgG fractions) from start of treatment to Day 15 | During the study from before administration of imlifidase up to Day 15
  Imlifidase cleaves IgG. PD of imlifidase will be assessed using a sodium dodecyl sulfate polyacrylamide gel electrophoresis (SDS-PAGE) analysis to measure the composition of the following fractions of IgG: Intact IgG, single cleaved IgG (scIgG) and Fab'2 fraction.
Anti-imlifidase antibody levels from start of imlifidase treatment to 6 months | During the study from before administration of imlifidase up to 6 months
  Only applicable for patients who receive imlifidase.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations, Study Director — Hansa Biopharma AB
Locations (48):
- United States (6):
  - UCLA Medical Center Plaza, Los Angeles, California
  - John Hopkins Medical Institution, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Minnesota Health Clinical Research Unit, Minneapolis, Minnesota
  - UNC Kidney Center/Division of Nephrology & Hypertension, Chapel Hill, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
- Austria (3):
  - Med Uni Graz / LKH-UNIV Klinikum Graz, Klinische Abteilung fuer Nephrologie, Graz, Stiermark
  - Medical University Innsbruck, Dept of Internal Medicine IV (Nephrology and Hypertension), Innsbruck, Tyrol
  - Medical University of Vienna, Dept of Medicine III, Division of Nephrology and dialysis, Vienna
- UZ Leuven, Leuven, Belgium
- Všeobecná fakultní nemocnice v Praze, Prague, Prague, Czechia
- Denmark (3):
  - Aarhus University Hospital, Renal Medicine and Clinical Medicine, Aarhus N, Central Jutland
  - Odense University Hospital, Medical Nephrology, Department Y, Odense, Region Syddanmark
  - Rigshospitalet, Department of Nephrology, Copenhagen
- France (9):
  - CHU Grenoble Alpes - Michallon Hospital, Nephrology, Hemodialysis, Apheresis and Kidney Transplantation, Grenoble, Auvergne-Rhône-Alpes
  - University Hospital of Marseille, Nephrology - Renal transplantation service, Marseille, Bouches-du-Rhône
  - Nouvel Hôpital Civil (University Hospital of Strasbourg), Strasbourg, Grand Est
  - CHU Lille. Nephrology, dialysis transplantation, Lille, Haus-de-France
  - CHU de Rouen, Department of Nephrology,Transplantation, and Hemodialysis, Bois-Guillaume, Normandy
  - CHU Bordeaux, Hôpital Pellegrin, Service nephrologie, transplantation, dialyse, aphereses, Bordeaux, Nouvelle-Aquitaine
  - Hôpital Rangueil, CHU de Toulouse, Department of Nephrology and Organ transplantation, Toulouse, Occitanie
  - CHU de Nantes, Hôtel-Dieu, Le service de néphrologie et immunologie clinique, Nantes, Pays de la Loire Region
  - Tenon Hospital, Renal intensive care unit, Paris, Île-de-France Region
- Germany (7):
  - LMU Klinikum, Medical Clinic IV / Department of Nephrology, Munich, Bavaria
  - Uniklinik RWTH Aachen, Aachen, North Rhine-Westphalia
  - Uniklinik Koeln-Klinik II fuer Innere Medizin, Cologne, North Rhine-Westphalia
  - Carl-Gustav-Carus University Hospital, Medizinische Klinik III, Nephrologie, Dresden, Saxony
  - Charité Department of Nephrology and Intensive Care, Berlin
  - Universitaetsklinikum Erlangen - Medizinische Klinik 4, Erlangen
  - University Hospital Hamburg-Eppendorf, III Department of Medicine and Nephrology, Hamburg
- Department of Renal Medicine, Cork University Hospital, Cork, Ireland
- Italy (3):
  - IRCCS Policlinico San Martino University Hospital, Department of Internal Medicine, Division of Nephrology, Genova, Genova-Liguria
  - IRCCS S. Orsola - Malpighi University Hospital - Nephrology, Dialysis and Transplantation Unit (pav 15), Bologna
  - ASST degli Spedali Civili di Brescia - SC Nefrologia, Brescia
- Netherlands (3):
  - Leiden University Medical Center, Department of Nephrology, Leiden, South Holland
  - University Medical Center Groningen, Division of Nephrology, Groningen
  - Radboudumc, Nijmegen
- Spain (2):
  - University Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
- Sweden (4):
  - Karolinska University Hospital, Huddinge
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Department of Nephrology, Lund
  - Uppsala University Hospital, Department of Medical Sciences, Renal Medicine, Uppsala
- United Kingdom (5):
  - Cambridge University Hospitals NHS Foundation Trust, Addenbrooke's Hospital, Dept. of Vasculitis, Cambridge, Cambridgeshire
  - Royal Infirmary of Edinburgh, Department of Renal Medicine, Edinburgh
  - University College London, Royal Free Hospital, Department of Renal Medicine, London
  - Hammersmith Hospital, Renal medicine and centre for inflammatory diseases, London
  - Manchester University Hospitals NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No